CLINICAL TRIAL: NCT00614107
Title: Organization in Acute Atrial Fibrillation Post Open Heart Surgery
Acronym: A-Fib
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Gregory Fink, SUNY Upstate Medical UNiversity
Other Study IDs: 5301UMU
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2008-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation post open heart surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue sample for the right and left sid eof the heart.
Oversight: Data Monitoring Committee: No

SUMMARY:
A form of irregular heart rate called, Atrial Fibrillation (AF) is a major clinical problem. It afflicts about 2 million Americans and is the single largest heart related cause of stroke. However, despite 120 years of speculation and research, the mechanisms that cause AF are poorly understood. Acute AF is also the most common irregular heart rate after open-heart surgery in patients. This is seen in as many as 30% of such patients and often results in a longer hospital stay.

In this study we would like to study the pattern of atrial fibrosis (scar tissue in the heart) and an associated blood marker (a protein called pro-collagen-1) in those patients concurrently having open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age, Male or Female
2. Able to provide consent
3. Cardiac surgery, CABG of Valve replacement or repair.

Exclusion Criteria:

1. If AF terminates within 1 hour of initiation.
2. If the patient undergoes electrical cardioversion and/or receives digitalis within the first hour of inclusion.
3. If the patients and/or their family or the primary caregiver choose to be excluded from the study anytime, even after the initial 24-hour period.
4. If the patient expires within 1 hour of inclusion into the study. -

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person over 18 years having an elective valve, CABG or combination procedure
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States